CLINICAL TRIAL: NCT06536673
Title: Educational Intervention Aimed At Reducing Infectious Complications Related to Peritoneal Dialysis
Brief Title: Intervention to Reduce Infectious Complications of Peritoneal Dialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Elena Fernandez Labadia, PhD student, Universitat de Lleida
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIC-2900
Record Dates: First submitted 2024-07-16; First posted 2024-08-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peritoneal Infection
Keywords: Educational intervention; Peritoneal dialysis; Peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Intervention Model Description: A retrospective control group with patients starting DP before January 2020 will be included and compared with an intervention group that will systematically include all patients starting DP since the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retrospective control group (Other): This is the PD population sample from before January 2020.
  Interventions: Behavioral: Data collection from the patient's clinical history
- Prospective study group (Experimental): It will be the incident patients in PD who will receive the educational intervention contained in this project and whose results will be compared with the control group.
  Interventions: Behavioral: Intervention to reduce infectious complications of peritoneal dialysis

INTERVENTIONS:
Behavioral: Intervention to reduce infectious complications of peritoneal dialysis — * Before catheter placement: The nurse and doctor provide the patient and/or caregiver with a PD simulation.
  * Initial training: from the placement of the catheter to the beginning of the technique at home, approximately 4 weeks, 6 and 7 sessions, duration 1-2 hours per session. Individualized learning taking into account learning abilities and education. It includes the explanation of the PD and the display of informational pictograms/capsules.
  * Step-by-step teaching: peritoneal exchange, peritoneal orifice care, administration of intraperitoneal medication, recording of constants, detection of complications and risk behaviors.
  * Nutritional education and water intake.
  * Administration of the Objective Structured Assessment (OSA) checklist.
  * Retraining: between the 1st and 3rd month of the start, after an episode of peritonitis and/or hospitalization, risk behaviors, functional/cognitive impairment, passivity/demotivation behaviors, and regularly once the year.
  Other Names: Prospective study group
  Arms: Prospective study group
Behavioral: Data collection from the patient's clinical history — Data collection from the patient's clinical history because this new standardized educational intervention was not used.
  Other Names: Retrospective control group
  Arms: Retrospective control group

SUMMARY:
Peritonitis is a common and serious complication of peritoneal dialysis (PD) and is one of the main causes of peritoneal dialysis technique failure and long-term hemodialysis conversion.

DETAILED DESCRIPTION:
Peritoneal infections (PI) have been a very relevant representative of peritoneal dialysis (PD) for decades. PI is a very serious complication of PD and is a source of concern because of its high incidence. Each episode carries clinical consequences for the patient, increases in treatment costs, hospital admissions, technical failures and risk of death, especially in the 30 days following an episode.

The risk of peritonitis depends on non-modifiable factors (such as age, sex, diabetes) and modifiable factors (such as anti-infective prophylaxis, catheter care, and training).

It is important to accurately analyze the effect of modifiable factors, as they are the most relevant in reducing the rate of peritonitis.

Patient education is very important and can affect the success of the technique and clinical results. Therapeutic education has been considered a key factor in PD outcomes.

The PD nurse is responsible for training the patient and/or caregiver to be self-sufficient and autonomous in care, reinforce and highlight the importance of adherence to treatment, and promote safe actions to prevent technique-related infections when this one is made at home.

This is a pragmatic, retrospective-prospective (ambispective) study of educational intervention for patients with stage V advanced chronic kidney disease and those with cardiorenal syndrome starting a peritoneal dialysis program.

A retrospective control group with patients starting PD before January 2020 will be included and compared with an intervention group that will systematically include all patients starting DP since the start of the study and they will be implemented a new educational intervention based on a systematic review that has been carried out with the most recent evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Medically stable
* Who can perform dialysis themselves or with the help of a caregiver willing to participate in the study and sign the informed consent will be included

Exclusion Criteria:

* Patients with psychiatric, psychological disorders and social (language barrier included)
* Who do not have a formal/informal caregiver
* Those who due to medical needs cannot continue with the standard schedule, pregnant women, participants who suffered peritonitis before receiving the educational intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of peritonitis | 1 year after educational intervention.
  It is calculated as the number of episodes of peritonitis per patient and year at risk.

SECONDARY OUTCOMES:
Age | Day 1 of peritoneal technique training.
  In years
Gender | Day 1 of peritoneal technique training.
  Male or female
Language barrier | Day 1 of peritoneal technique training.
  Yes or not
Marital status | Day 1 of peritoneal technique training.
  Single, married, coupled, separated - divorced, widowed
Educational level | Day 1 of peritoneal technique training.
  Not finished primary studies, primary schools, secondary, middle/higher grade cycle, high school, university studies, doctorate
Caregiver disposition | Day 1 of peritoneal technique training.
  Yes or not
Drinking water supply | Day 1 of peritoneal technique training.
  Yes or not
Weight | Day 1 of peritoneal technique training.
  In kilograms
Height | Day 1 of peritoneal technique training.
  In meters
Body Mass Index (BMI) | Day 1 of peritoneal technique training.
  BMI= Current weight (kg) ÷ height (m) x height (m)= kg/m2. Low weight: Less than 18.4 Normal weight: 18.5 to 24.9 Overweight: 25 to 29.9 Grade I Obesity: 30 to 34.9 Grade II Obesity: 35 to 39.9 Grade III Obesity: Equal to or greater than 40.
Diabetes | Day 1 of peritoneal technique training.
  Yes or not
Cardiovascular disease | Day 1 of peritoneal technique training.
  Yes or not
Cerebrovascular disease | Day 1 of peritoneal technique training.
  Yes or not
Hypertension | Day 1 of peritoneal technique training.
  Yes or not
Cancer | Day 1 of peritoneal technique training.
  Yes or not
The primary cause of kidney disease | Day 1 of peritoneal technique training.
  Glomerular disease, tubulointerstitial disease, diabetes mellitus, hypertension, other systemic diseases, familial/hereditary nephropathy, various renal disorders
Barthel index | Day 1 of peritoneal technique training.
  Scores of 100 imply total independence. Scores between 100 and 60 indicate the existence of a slight dependency or need for help, between 55 and 40 a moderate dependency, from 35 to 20 we would speak of severe dependency and scores below 20 points would indicate that the subject has a total dependence
Lawton and Brody scale | Day 1 of peritoneal technique training.
  The 8 points indicate total independence to carry out the instrumental activities of daily life.- A lower result indicates functional deterioration.
Assessment of quality of life with the questionnaire EuroQol-5D (EQ-5D) | Day 1 of peritoneal technique training.
  They are coded as 1 if the response option is "I have no problems"; with a 2 if the response option is "some or moderate problems"; and with a 3 if the answer option is "many problems." In such a way that the higher the value reflected, the worse the assessment that the subject makes of his or her state.
Cognitive impairment -PFEIFFER Test | Day 1 of peritoneal technique training.
  From 0 to 2 errors: The patient is considered to have no cognitive impairment. 3 to 4 errors: The patient is considered to have mild cognitive impairment. From 5 to 7 errors: The patient is considered to have moderate cognitive impairment
Fragility detection - Q-Scale FRAIL | Day 1 of peritoneal technique training.
  Between 1-2 affirmative answers: pre-fragile. >2 fragile
The origin before arriving at peritoneal dialysis | Day 1 of peritoneal technique training.
  Pre-dialysis, hemodialysis, transplantation, cardiorenal syndrome
Residual renal function | Day 1 of peritoneal technique training.
  Yes or not
Type of peritoneal catheter | Day 1 of peritoneal technique training.
  Self-positioning catheter/Tenckhoff straight
Hemoglobin | First month of the start of the technique at home.
  12.0 - 16.0 gr/dl
Serum albumin | First month of the start of the technique at home.
  3.4 - 5.2 g/dL
Serum potassium | First month of the start of the technique at home.
  3.50 - 5.50 mmol/L
Serum sodium | First month of the start of the technique at home.
  135.0 - 150.0 mmol/L
Serum bicarbonate | First month of the start of the technique at home.
  23.0 - 27.0 mmol/L
Serum calcium | First month of the start of the technique at home.
  8.80 - 10.60 mg/dL
Serum phosphorus | First month of the start of the technique at home.
  2.70 - 4.50 mg/dL
Blood urea nitrogen | First month of the start of the technique at home.
  10 - 50 mg/dL
Serum creatinine | First month of the start of the technique at home.
  0.50 - 0.90 mg/dL
Peritonitis | Follow-up during the first year after educational intervention.
  Yes or not
Time to first peritonitis | Follow-up during the first year after educational intervention.
  In months without peritonitis
Orifice infection | Follow-up during the first year after educational intervention.
  Yes or not
Peritoneal orifice tunnelitis | Follow-up during the first year after educational intervention.
  Yes or not
Result of peritoneal fluid culture | Follow-up during the first year after educational intervention.
  positive, negative
Type of peritoneal infection | Follow-up during the first year after educational intervention.
  Germ, fungus, biofilm
Reinfection | Follow-up during the first year after educational intervention.
  Yes or not
Relapse | Follow-up during the first year after educational intervention.
  Yes or not
Complicated peritonitis | Follow-up during the first year after educational intervention.
  change of technique/death
Antibiotic administered | Follow-up during the first year after educational intervention.
  Type of antibiotic administered, the dosage.

REFERENCES:
- [Background] Bonnal H, Bechade C, Boyer A, Lobbedez T, Guillouet S, Verger C, Ficheux M, Lanot A. Effects of educational practices on the peritonitis risk in peritoneal dialysis: a retrospective cohort study with data from the French peritoneal Dialysis registry (RDPLF). BMC Nephrol. 2020 May 29;21(1):205. doi: 10.1186/s12882-020-01867-w. PMID 32471380
- [Background] Cho Y, Htay H, Johnson DW. Centre effects and peritoneal dialysis-related peritonitis. Nephrol Dial Transplant. 2017 Jun 1;32(6):913-915. doi: 10.1093/ndt/gfx054. No abstract available. PMID 28505351
- [Background] Gadola L, Poggi C, Poggio M, Saez L, Ferrari A, Romero J, Fumero S, Ghelfi G, Chifflet L, Borges PL. Using a multidisciplinary training program to reduce peritonitis in peritoneal dialysis patients. Perit Dial Int. 2013 Jan-Feb;33(1):38-45. doi: 10.3747/pdi.2011.00109. Epub 2012 Jul 1. PMID 22753455
- [Background] Bieber S, Mehrotra R. Peritoneal Dialysis Access Associated Infections. Adv Chronic Kidney Dis. 2019 Jan;26(1):23-29. doi: 10.1053/j.ackd.2018.09.002. PMID 30876613
- See also: Clinical guide of the Spanish Society of Nephrology on the prevention and treatment of peritoneal infection in peritoneal dialysis — https://doi.org/10.1016/J.NEFRO.2021.10.007